CLINICAL TRIAL: NCT05426785
Title: A Multicenter Prospective Randomized Study to Evaluate the Delivery Timing Safety and Efficacy of AntiTachycardia Pacing
Brief Title: To Evaluate the Delivery Timing Safety and Efficacy of AntiTachycardia Pacing (BIO|ATP)
Acronym: BIO|ATP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Collaborators: Biotronik Japan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA119
Record Dates: First submitted 2022-06-07; First posted 2022-06-22 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Implantable Cardioverter Defibrillator(ICD)
Keywords: ICD; shock; Antitachycardiac Pacing(ATP); Ventricular Tachycardia(VT); Ventricular Fibrillation(VF); Ventricular arrhythmias(VA)
MeSH Terms: conditions — Shock; Tachycardia, Ventricular; Ventricular Fibrillation | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group(Early Multiple ATP Group) (Active Comparator): Set to perform multiple ATP early
  Interventions: Device: 1:1 ratio for Treatment Group and Control Group
- Control Group (Active Comparator): Set the extended detection time for the conventional ATP (Refer to the settings of "Delayed Therapy-arm C" in Multicenter Automatic Defibrillator Implantation Trial - Reduce Inappropriate Therapy (MADIT-RIT) study)
  Interventions: Device: 1:1 ratio for Treatment Group and Control Group

INTERVENTIONS:
Device: 1:1 ratio for Treatment Group and Control Group — Randomization also will be performed at latest 10 days after ICD implantation, and the specified device programming settings for the allocated group will be set after successful implantation of the investigational devices.

SUMMARY:
To compare Treatment Group (settings of Early Multiple ATP) and Control Group (settings of extended detection time for the conventional ATP) in Japanese patients, and confirm their safety and efficacy

DETAILED DESCRIPTION:
The enrolled patients are randomized to Treatment Group with setting to provide Antitachycardiac Pacing (ATP) multiple times at an early timing or Control Group with Long Detection setting for the conventional ATP, at latest 10 days after the implantation of the Implantable Cardioverter Defibrillator(ICD) system in the domestic centers to confirm the safety and efficacy of the setting for the early timing multiple ATP treatment in Japanese patients.

The follow-up is not pre-defined and the data (including the home monitoring data) is collected according to the site's standard outpatient schedule, but the data will be collected at the hospital visit for the initial appropriate or inappropriate shock therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient has an indication for ICD according to the The Japanese Circulation Society (JCS )/ Japanese Heart Rhythm Society (JHRS) 2021 Guideline Focused Update on Non-Pharmacotherapy of Cardiac Arrhythmias
* Patient is either planned for de novo ICD implantation or is already implanted with an investigational ICD for 10 days or less.
* Patient can be treated with ATP therapy for both VT and VF zone
* Patient is willing and able to use the CardioMessenger and accepts the Home Monitoring concept
* Patient is willing to visit the hospital in accordance with physician's instruction
* Patient is able to understand the nature of the study and to provide written informed consent

Exclusion Criteria:

* Patient planned for implantation with or already implanted with Cardiac Resynchronization Therapy Defibrillator (CRT-D) device
* A patient who is confirmed to have received ICD therapy
* A patient who is diagnosed as Idiopathic VF (e.g. Brugada syndrome, Long QT Syndrome, other IVF)
* Age < 18 years
* A patient who has impaired mental status
* Life expectancy less than 18 months
* Participation in another interventional clinical investigation
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Time to first shock by Kaplan-Meier approach | From a minimum of 18 months to a maximum of 42 months
  During the study duration(42 months: the enrollment period is 24 months plus the follow up period is 18 months from the Last Patient In(LPI)), to confirm that Treatment Group is the non-inferiority to the Control Group in terms of the time from randomized prescriptive settings to first shock with ICD device treatment, by Kaplan-Meier approach. The time frame of event evaluation is from a minimum of 18 months to a maximum of 42 months, since the study duration for each subject will differ according to the timing of enrollment.

SECONDARY OUTCOMES:
Success rate of the ATP | From a minimum of 18 months to a maximum of 42 months
  During the study duration (42 months: the enrollment period is 24 months plus the follow up period is 18 months from the Last Patient In(LPI)), calculate the percentage of successful ATP treatment for all collected ATP treatment episodes. The definition of ATP success is that confirming by one beat of sinus rhythm or Atrial Pacing (in case of Atrial fibrillation, the electrical complex on an Electrocardiogram (ECG) related to the depolarization of the ventricles (QRS) or Ventricular Pacing) under the tachycardia detection rate. The time frame of event collections is from a minimum of 18 months to a maximum of 42 months, since the study duration for each subject will differ according to the timing of enrollment.
Duration until the end of the episode | From a minimum of 18 months to a maximum of 42 months
  For all episodes collected during the study duration (42 months: the enrollment period is 24 months plus the follow up period is 18 months from the Last Patient In(LPI)), the time from the onset to the termination of the episode recorded in the ICD device is measured as the episode duration. The time frame of event collections is from a minimum of 18 months to a maximum of 42 months, since the study duration for each subject will differ according to the timing of enrollment.
Cardiac mortality | From a minimum of 18 months to a maximum of 42 months
  During the study duration (42 months: the enrollment period is 24 months plus the follow up period is 18 months from the Last Patient In(LPI)), confirm the occurrence of cardiac mortality in all enrolled patients.The time frame of evaluation of cardiac mortality is from a minimum of 18 months to a maximum of 42 months, since the study duration for each subject will differ according to the timing of enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Kenji Ando, Principal Investigator — Kokura Memorial Hospital
Locations (1):
- Kokura Memorial Hospital, Kitakyushu, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
The study is the domestic multicenter clinical study, and the Publication Steering Committee(PSC) consisting of researchers may perform the analysis in accordance with the decision by PSC after first publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after 6 months of Lst Patient Out (LPO)
Access Criteria: Following Sponsor'ｓStandard Operating Procedures ()

REFERENCES:
- [Result] Schuger C, Daubert JP, Zareba W, Rosero S, Yong P, McNitt S, Kutyifa V. Reassessing the role of antitachycardia pacing in fast ventricular arrhythmias in primary prevention implantable cardioverter-defibrillator recipients: Results from MADIT-RIT. Heart Rhythm. 2021 Mar;18(3):399-403. doi: 10.1016/j.hrthm.2020.11.019. Epub 2020 Nov 21. PMID 33232811
- [Result] Arenal A, Proclemer A, Kloppe A, Lunati M, Martinez Ferrer JB, Hersi A, Gulaj M, Wijffels MC, Santi E, Manotta L, Mangoni L, Gasparini M. Different impact of long-detection interval and anti-tachycardia pacing in reducing unnecessary shocks: data from the ADVANCE III trial. Europace. 2016 Nov;18(11):1719-1725. doi: 10.1093/europace/euw032. Epub 2016 Aug 2. PMID 27485577
- [Result] Sterns LD, Meine M, Kurita T, Meijer A, Auricchio A, Ando K, Leng CT, Okumura K, Sapp JL, Brown ML, Lexcen DR, Gerritse B, Schloss EJ. Extended detection time to reduce shocks is safe in secondary prevention patients: The secondary prevention substudy of PainFree SST. Heart Rhythm. 2016 Jul;13(7):1489-96. doi: 10.1016/j.hrthm.2016.03.022. Epub 2016 Mar 14. PMID 26988379
- [Result] Joung B, Lexcen DR, Ching CK, Silver MT, Piccini JP, Sterns LD, Rabinovich R, Pickett RA, Liu S, Brown ML, Cheng A. Additional antitachycardia pacing programming strategies further reduce unnecessary implantable cardioverter-defibrillator shocks. Heart Rhythm. 2020 Jan;17(1):98-105. doi: 10.1016/j.hrthm.2019.07.027. Epub 2019 Jul 29. PMID 31369873
- [Result] Yokoshiki H, Shimizu A, Mitsuhashi T, Ishibashi K, Kabutoya T, Yoshiga Y, Kohno R, Abe H, Nogami A; Members of the Implantable Cardioverter-Defibrillator (ICD) Committee of the Japanese Heart Rhythm Society. Trends in the use of implantable cardioverter-defibrillator and cardiac resynchronization therapy device in advancing age: Analysis of the Japan cardiac device treatment registry database. J Arrhythm. 2020 Jun 8;36(4):737-745. doi: 10.1002/joa3.12377. eCollection 2020 Aug. PMID 32782648